CLINICAL TRIAL: NCT03268369
Title: PET Study of the Nicotinic System in Epilepsy
Acronym: NICOPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabienne PICARD (Other)
Responsible Party: Sponsor-Investigator, Fabienne PICARD, Doctor, University Hospital, Geneva, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-041
Record Dates: First submitted 2017-08-24; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Active Comparator)
  Interventions: Radiation: MRI of the brain; Radiation: PET scan [18F]F-A-85380; Radiation: PET scan [18F]FDG
- Non lesional diurnal partial epilepsy (Experimental)
  Interventions: Radiation: MRI of the brain; Radiation: PET scan [18F]F-A-85380; Radiation: PET scan [18F]FDG
- Idiopathic generalized epilepsy (Experimental)
  Interventions: Radiation: MRI of the brain; Radiation: PET scan [18F]F-A-85380; Radiation: PET scan [18F]FDG
- Nocturnal frontal lobe epilepsy (Experimental)
  Interventions: Radiation: MRI of the brain; Radiation: PET scan [18F]F-A-85380; Radiation: PET scan [18F]FDG
- Epileptic patients with Vagus Nerve Stimulation (VNS) (Experimental)
  Interventions: Radiation: PET scan [18F]F-A-85380; Radiation: PET scan [18F]FDG

INTERVENTIONS:
Radiation: MRI of the brain — to eliminate a structural intra-cerebral lesion
  Arms: Control group; Idiopathic generalized epilepsy; Nocturnal frontal lobe epilepsy; Non lesional diurnal partial epilepsy
Radiation: PET scan [18F]F-A-85380 — exam performed after iv injection of 200 MBq [18F]F-A-85380
Radiation: PET scan [18F]FDG — exam performed after iv injection of 200 MBq [18F]FDG

SUMMARY:
Mutations in neuronal nicotinic acetylcholine receptors (nAChRs) have been identified in the autosomal dominant nocturnal frontal lobe epilepsy (ADNFLE). Despite the demonstration of a gain of function of the mutated receptors, the precise mechanisms leading to this nocturnal epilepsy are still unknown. In 2006 the investigators studied the nAChR cerebral distribution in a group of patients with ADNFLE carrying a nAChR mutation, by a PET-scan using [18F]-F-A-85380, a ligand with a high affinity and specificity for alpha4beta2 nicotinic receptors. The study showed a different pattern of brain distribution of the radiotracer in the ADNFLE patients when compared to a group of control subjects, with a significant increase of nicotinic receptor density in the patients in mesencephalon and cerebellum (Picard et al., Brain 2006). Based on the known biochemical and cellular circuits in the brainstem, these results suggest that the nAChR density increase in mesencephalon is involved in the pathophysiology of ADNFLE through the role of brainstem ascending cholinergic systems in arousal. The follow-up step consists of extending this examination to other forms of epilepsy, in order to verify the specificity of the hyperfixation pattern for ADNFLE, and search for a potential involvement of nicotinic receptors in other forms of epilepsy. The investigators aim to study 5 groups of subjects: control subjects (Group 1, 20 subjects); patients with a non lesional partial epilepsy and a predominance of diurnal seizures (Group 2, 12 subjects); patients with an idiopathic generalized epilepsy (Group 3, 12 subjects); patients with nocturnal frontal lobe epilepsy (Group 4, 3 subjects) and epileptic patients with vagal nerve stimulation (Group 5, 1 subject). For each patient, a cerebral MRI, [18F]- fluorodeoxyglucose (FDG) PET/CT and [18F]-F-A-85380 PET/CT examinations are planned. The investigators will perform data analyses on volume of distribution (Vt) parametric images which will be based on the ratio of brain tissue to unchanged F-A-85380 plasma at equilibrium. Statistical parametric mapping (SPM2) will be used to further study the parametric PET images. This study is primarily dedicated to demonstrate that the pattern of hyperfixation that was obtained in ADNFLE patients is specific for this disorder and does not constitute a common pattern to various forms of epilepsy. The investigators will also search for a possible involvement of the nAChRs in other forms of epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* males
* 18-60 years old
* non-smokers

Exclusion Criteria:

* smoking during the past twelve months
* contraindications to MRI
* brain lesions on MRI (including hippocampal atrophy)
* neurological disorder (other than epilepsy) or psychiatric disorder
* neoplasia or coronary disease
* blood test showing : creatinine clearance < 50 ml/min, or platelet < 100 G/l, or leucocytes < 3.8 G/l, or ALT or AST > 2 x upper standard, or gamma-GT > 3 x upper standard, or albumin < 35 g/l or > 48 g/l .
* patients only : nuclear imaging during the past twelve months
* healthy volunteers only : ionising radiation exam during the past five years

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the cerebral distribution of the neuronal nicotinic acetylcholine receptors (nAChR) in the 5 groups of individuals by means of voxelwise and regional 18F-FA binding potential measurements | 1 month
  Parametric 18F-FA and 18F-FDG binding potential measurements will be compared between the different groups of patients with epilepsy and the control group in order to find specific changes in the cerebral distribution of the nicotinic receptors in the different types of epilepsy, by using a voxel-wise (SPM) and a volume of interest (VOI) analysis.

REFERENCES:
- [Background] Picard F, Bruel D, Servent D, Saba W, Fruchart-Gaillard C, Schollhorn-Peyronneau MA, Roumenov D, Brodtkorb E, Zuberi S, Gambardella A, Steinborn B, Hufnagel A, Valette H, Bottlaender M. Alteration of the in vivo nicotinic receptor density in ADNFLE patients: a PET study. Brain. 2006 Aug;129(Pt 8):2047-60. doi: 10.1093/brain/awl156. Epub 2006 Jun 30. PMID 16815873